CLINICAL TRIAL: NCT04603469
Title: Incidence of Hypotension in Children With Down Syndrome During Induction of Anesthesia With Sevoflurane
Brief Title: Hypotension in Children With Down Syndrome With Anesthesia Induction
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Adam Adler MD, MS, FAAP, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-48044
Record Dates: First submitted 2020-10-21; First posted 2020-10-26 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Hypotension on Induction
MeSH Terms: interventions — Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trisomy 21 patients: Children <18 years old requiring general anesthesia with inhalation induction Down syndrome ASA physical classification 1-3
  Interventions: Other: Non invasive blood pressure

INTERVENTIONS:
Other: Non invasive blood pressure — measurement of blood pressure during induction of general anesthesia
  Other Names: blood pressure

SUMMARY:
Children generally undergo induction of anesthesia by inhalation of sevoflurane. Children with Down Syndrome experience bradycardia with induction of anesthesia using sevoflurane. It is unknown if this bradycardia is isolate or results in hypotension, thus requiring treatment. Isolate bradycardia without hypotension does not require treatment and should be avoided as many of these patients have underlying cardiac anomalies.

DETAILED DESCRIPTION:
Children generally undergo induction of anesthesia by inhalation of sevoflurane. This is particularly relevant for children with developmental delays as to avoid placement of an IV while awake. However, children with Down Syndrome experience bradycardia with induction of anesthesia using sevoflurane. It is unknown if this bradycardia is isolate or results in hypotension, thus requiring treatment. Isolate bradycardia without hypotension does not require treatment and should be avoided as many of these patients have underlying cardiac anomalies.

ELIGIBILITY:
Inclusion Criteria:

Children <18 years old Requiring general anesthesia with inhalation induction Down syndrome ASA physical classification 1-3

Exclusion Criteria:

Patients >18 years of age Patients without down syndrome Cyanotic congenital heart disease Use of antihypertensive medications Pulmonary hypertension patients undergoing intravenous induction of anesthesia ASA physical classification other than 1-3 emergency procedure

Ages: 1 Week to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This is an observational study of children with down syndrome undergoing induction of general anesthesia with sevoflurane. vital signs of blood pressure, heart rate and pulse oximetry will be recorded on the anesthesia record as standard practice
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Assessment of non-invasive blood pressure during induction | 5 minutes
  non invasive blood pressure during induction (systolic, diastolic and Mean pressures)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Adler, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Childrens Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No